CLINICAL TRIAL: NCT00317408
Title: Treatment Protocol for Relapsed Anaplastic Large Cell Lymphoma of Childhood and Adolescence
Brief Title: Combination Chemotherapy Followed By Stem Cell Transplant in Treating Young Patients With Progressive or Relapsed Anaplastic Large Cell Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Inter-group Cooperation on Childhood and Adolescent Non Hodgkin Lymphoma (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000466639; EICNHL-ALCL-RELAPSE; AIEOP-EICNHL-ALCL-RELAPSE; BFM-EICNHL-ALCL-RELAPSE; BSPHO-EICNHL-ALCL-RELAPSE; DCOG-EICNHL-ALCL-RELAPSE; NOPHO-EICNHL-ALCL-RELAPSE; PPLLSG-EICNHL-ALCL-RELAPSE; SFCE-EICNHL-ALCL-RELAPSE; SHOP-EICNHL-ALCL-RELAPSE; CCLG-NHL-2006-01; EU-205118; EU-20618; EUDRACT-2005-003321-57
Record Dates: First submitted 2006-04-19; First posted 2006-04-24 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Lymphoma
Keywords: anaplastic large cell lymphoma; recurrent childhood anaplastic large cell lymphoma; stage III childhood anaplastic large cell lymphoma; stage IV childhood anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic | interventions — Antilymphocyte Serum; Busulfan; Carboplatin; Carmustine; Cyclosporine; Cytarabine; Dexamethasone; etoposide phosphate; Idarubicin; Ifosfamide; Leucovorin; Lomustine; Melphalan; Methotrexate; Mitoxantrone; Prednisolone; Thiotepa; Vinblastine; Vindesine; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: carboplatin
Drug: carmustine
Drug: cyclosporine
Drug: cytarabine
Drug: dexamethasone
Drug: etoposide phosphate
Drug: idarubicin
Drug: ifosfamide
Drug: leucovorin calcium
Drug: lomustine
Drug: melphalan
Drug: methotrexate
Drug: mitoxantrone hydrochloride
Drug: prednisolone
Drug: thiotepa
Drug: vinblastine sulfate
Drug: vindesine
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: autologous hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Giving combination chemotherapy and total-body irradiation before a peripheral stem cell transplant that uses the patient's or a donor's stem cells, helps stop both the growth of cancer cells and the patient's immune system from rejecting the stem cells. When the stem cells are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Giving combination chemotherapy and total-body irradiation followed by a stem cell transplant may be an effective treatment for anaplastic large cell lymphoma.

PURPOSE: This clinical trial is studying how well combination chemotherapy followed by stem cell transplant works in treating young patients with progressive or relapsed anaplastic large cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Improve the probability of event-free survival in children and adolescents with early progression of anaplastic large cell lymphoma (ALCL) and/or relapse of ALCL with CD3-positive immunophenotype treated with reinduction combination chemotherapy followed by allogeneic or autologous stem cell transplantation.
* Determine whether a conditioning regimen comprising carmustine, etoposide phosphate, cytarabine, and melphalan (BEAM) (without total body irradiation) for autologous stem cell transplantation is an effective treatment for patients with relapsed CD3-negative ALCL occurring after the intensive phase of treatment.
* Determine the impact of vinblastine in patients with late relapse of CD3-negative ALCL who have not received vinblastine during frontline therapy.

Secondary

* Determine overall survival and treatment-related mortality in patients treated with these regimens.
* Determine acute and long-term toxicity in patients treated with these regimens.
* Determine the rate of acute and chronic graft-vs-host disease in patients treated with allogeneic stem cell transplantation.

OUTLINE: This is a multicenter, prospective, nonrandomized study. Patients are stratified according to time from initial diagnosis to progression/relapse, immunophenotype of lymphoma cells (CD3-positive + vs CD3-negative), stem cell donor availability (matched sibling donor vs 9/10 or 10/10 matched unrelated donor), and vinblastine during frontline therapy (yes vs no).

* Group 1 (early progression): Patients receive 1 course of ICM chemotherapy followed by 1 course of ICI chemotherapy.

  * ICM chemotherapy: Patients receive methotrexate, cytarabine, and prednisolone intrathecally (IT) on day 1, mitoxantrone hydrochloride IV over 5 hours on days 1 and 2, carboplatin IV continuously on days 2-5 and ifosfamide IV continuously on days 2-6.
  * ICI chemotherapy: Patients receive methotrexate, cytarabine, and prednisolone intrathecally on day 1, idarubicin IV over 4 hours on days 1 and 2, carboplatin IV continuously on days 2-5, and ifosfamide IV continuously on days 2-6.

Patients then proceed to allogeneic stem cell transplantation.

* Group 2 (relapsed disease and CD3-positive lymphoma cells): Patients are stratified according to stem cell donor availability (yes vs no).

  * Available donor: Patients receive 2 courses of CC chemotherapy and then proceed to allogeneic stem cell transplantation.
  * Unavailable donor : Patients receive 2 courses of CC chemotherapy comprising dexamethasone orally or IV on days 1-5, vindesine IV on day 1, cytarabine IV over 3 hours on days 1 and 2, etoposide phosphate IV over 2 hours on days 3-5, and methotrexate, cytarabine, and prednisolone IT on day 5. Patients then receive 1 course of CVA chemotherapy comprising oral lomustine on day 1, vinblastine IV on days 1, 8, 15, and 22, and cytarabine IV over 1 hour on days 1-5. Patients undergo leukapheresis for collection of autologous peripheral blood stem cells after the first and/or second course of CC chemotherapy. Patients then proceed to autologous stem cell transplantation.
* Group 3 (relapsed disease, CD3-negative immunophenotype, and received vinblastine during frontline therapy): Patients receive 2 courses of CC chemotherapy and 1 course of CVA chemotherapy as described above. Patients undergo leukapheresis for collection of autologous peripheral blood stem cells (PBSC) after the first and/or second course of CC chemotherapy. Patients then proceed to autologous stem cell transplantation.
* Group 4 (late relapse, CD3-negative immunophenotype, and did not receive vinblastine during frontline therapy): Patients receive vinblastine IV once weekly for 24 months. Patients with disease progression during or relapsed disease after vinblastine therapy undergo treatment as in group 3.
* Autologous stem cell transplantation (SCT): Patients receive a conditioning regimen comprising carmustine IV over 1 hour on day -7, etoposide phosphate IV over 1 hour and cytarabine IV over 30 minutes on days -6 to -3, and melphalan IV over 15 minutes on day -2. Patients undergo autologous SCT on day 0.
* Allogeneic SCT: Beginning 4-6 weeks after the start of the last chemotherapy course, patients receive 1 of the following conditioning regimens based on age:

  * Patients > 2 years of age undergo total body irradiation on days -7 to -5 and receive thiotepa IV over 1 hour on day -4 and etoposide IV over 4 hours on day -3. Patients undergo allogeneic SCT on day 0.
  * Patients ≤ 2 years of age receive oral busulfan 4 times daily on days -8 to -5, thiotepa IV over 1 hour twice on day -4, and etoposide phosphate IV over 4 hours on day -3. Patients undergo allogeneic SCT on day 0.

Patients undergoing SCT from an unrelated donor also receive antithymocyte globulin IV over 4 hours on days -3 to -1.

All patients receive graft-versus-host (GVHD) prophylaxis as described below.

* GVHD prophylaxis: GVHD prophylaxis is administered as per donor status.

  * Matched sibling donor: Patients receive cyclosporine IV over 2 hours or orally on day -1 to 60 followed by a taper.
  * 10/10 or 9/10 matched unrelated donor: Patients receive cyclosporine IV over 2 hours or orally on days -1 to 100 followed by a taper, methotrexate IV on days 1, 3, and 6, and leucovorin calcium IV on days 2, 4, and 7.
  * Mismatched donor: Patients do not receive GVHD prophylaxis, however, CD3-positive lymphocytes are extracted from donor stem cells.

After completion of study treatment, patients are followed periodically for 10 years.

PROJECTED ACCRUAL: A total of 96 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed anaplastic large cell lymphoma (ALCL)

  * Progressive disease OR first relapse
  * No second or subsequent relapse of ALCL
* Slides available for national central pathology review
* Availability of 1 of the following (for allogeneic stem cell transplantation only):

  * HLA-identical matched sibling donor
  * 10/10 HLA-matched nonsibling donor (related or unrelated)
  * 9/10 HLA-matched nonsibling donor (1-antigen-mismatched related or unrelated donor)
  * < 9/10 HLA-mismatched donor (related or unrelated)

    * Stem cells may be obtained from unmanipulated bone marrow or peripheral blood stem cells after filgrastim (G-CSF) stimulation

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Adequate hepatic, renal, and cardiac function
* No HIV infection or AIDS
* No severe immunodeficiency
* No other prior malignancy
* No pre-existing disease or condition prohibiting study treatment

PRIOR CONCURRENT THERAPY:

* At least 2 months since prior chemotherapy or radiotherapy
* No significant pretreatment for first relapse
* No prior organ transplantation
* No concurrent participation in another clinical trial

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2004-04; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Event-free survival as measured by the Kaplan-Meier method

SECONDARY OUTCOMES:
Proportion of patients who are treated on protocol among all patients who meet the inclusion criteria
Overall survival
Acute and long term toxicity
Rate of acute and chronic graft-vs-host disease in patients with allogeneic stem cell transplantation
Treatment related mortality

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Reiter, MD, Study Chair — University Hospital Erlangen; Denise Williams, MD — Cambridge University Hospitals NHS Foundation Trust
Locations (98):
- St. Anna Children's Hospital, Vienna, Austria
- U.Z. Gasthuisberg, Leuven, Belgium
- Czechia (2):
  - University Hospital Brno, Brno
  - Charles University Hospital, Prague
- Centre Leon Berard, Lyon, France
- Germany (62):
  - Kinderklinik - Universitaetsklinikum Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Helios Klinikum Berlin, Berlin
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Evangelisches Krankenhauus Bielfeld, Biefeld
  - Kinderklinik der Universitaet Bonn, Bonn
  - Staedtisches Klinikum - Howedestrase, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Kliniken der Stadt Koeln gGmbH - Kinderkrankenhaus Riehl, Cologne
  - Children's Hospital, Cologne
  - Carl - Thiem - Klinkum Cottbus, Cottbus
  - Vestische Kinderklinik, Datteln
  - Klinikum Dortmund, Dortmund
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Helios Klinikum Erfurt, Erfurt
  - Universitaets - Kinderklinik, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitaetskinderklinik - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Kinderklinik, Giessen
  - Universitaetsklinikum Goettingen, Göttingen
  - Klinik und Poliklinik Fuer Kinder-und Jugendmedizin - Universitaetsklinikum Greifswald, Greifswald
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaets-Kinderklinik Heidelberg, Heidelberg
  - Gemeinschaftskrankenhaus, Herdecke
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitaets - Kinderklinik, Jena
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Klinikum Kassel, Kassel
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Klinikum Kemperhof Koblenz, Koblenz
  - Klinikum Krefeld GmbH, Krefeld
  - Universitaets - Kinderklinik, Leipzig
  - St. Annastift Krankenhaus, Ludwigshafen
  - Universitaets - Kinderklinik - Luebeck, Lübeck
  - Universitatsklinikum der MA, Magdeburg
  - Johannes Gutenberg University, Mainz
  - Staedtisches Klinik - Kinderklinik, Mannheim
  - Universitaets - Kinderklinik, Marburg
  - Klinikum Minden, Minden
  - Krankenhaus Muenchen Schwabing, Munich
  - Dr. von Haunersches Kinderspital der Universitaet Muenchen, Munich
  - Klinik und Poliklinik fuer Kinder und Jugendmedizin - Universitaetsklinikum Muenster, Münster
  - Kinderklinik Kohlhof, Neunkirchen
  - Cnopf'sche Kinderklinik, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - Klinik St. Hedwig-Kinderklinik, Regensburg
  - Kinderklinik - Universitaetsklinikum Rostock, Rostock
  - Saarbrucker Winterbergkliniken, Saarbrücken
  - Johanniter-Kinderklinik, Sankt Augustin
  - Klinikum Schwerin, Schwerin
  - Kinderklink Siegen Deutsches Rotes Kreuz, Siegen
  - Olgahospital, Stuttgart
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Universitaetsklinikum Tuebingen, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Helios Kliniken Wuppertal University Hospital, Wuppertal
  - Universitaets - Kinderklinik Wuerzburg, Würzburg
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- Azienda Ospedaliera di Padova, Padua, Italy
- Erasmus MC - Sophia Children's Hospital, Rotterdam, Netherlands
- Akademia Medyczna im. Piastow Slaskich, Wroclaw, Poland
- Goeteborg University, Gothenburg, Sweden
- Switzerland (6):
  - Kantonspital Aarau, Aarau
  - Universitaets-Kinderspital beider Basel, Basel
  - Ospedale "la Carita", Locarno, Locarno
  - Kinderspital Luzern, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - University Children's Hospital, Zurich
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Middlesex Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales

REFERENCES:
- [Derived] Knorr F, Zimmermann M, Bader P, Lang P, Muller I, Basu O, Burkhardt B, Seidl J, Damm-Welk C, Pichler H, Attarbaschi A, Meissner B, Beier R, Woessmann W. Allogeneic HSCT for consolidation in pediatric refractory or relapsed ALK-positive anaplastic large cell lymphoma. Blood Adv. 2026 Feb 3:bloodadvances.2025018774. doi: 10.1182/bloodadvances.2025018774. Online ahead of print. PMID 41632689
- [Derived] Knorr F, Brugieres L, Pillon M, Zimmermann M, Ruf S, Attarbaschi A, Mellgren K, Burke GAA, Uyttebroeck A, Wrobel G, Beishuizen A, Aladjidi N, Reiter A, Woessmann W; European Inter-Group for Childhood Non-Hodgkin Lymphoma. Stem Cell Transplantation and Vinblastine Monotherapy for Relapsed Pediatric Anaplastic Large Cell Lymphoma: Results of the International, Prospective ALCL-Relapse Trial. J Clin Oncol. 2020 Dec 1;38(34):3999-4009. doi: 10.1200/JCO.20.00157. Epub 2020 Jul 30. PMID 32730187